CLINICAL TRIAL: NCT07379892
Title: Evaluatıon of TREM-1, MMP-8 and TIMP-1 Levels in Perı-Implant Crevicular Fluıd of Perı-Implanted Indıvıduals
Status: Completed | Type: Observational
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, Veli Özgen Öztürk, Principal Investigator, Aydin Adnan Menderes University
Other Study IDs: BAP-23003
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Periimplantitis
Keywords: periimplantitis; TREM-1; MMP-8; TIMP-1
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Peri-implantitis: Peri-implantitis is defined as bleeding on probing, suppuration, increased probing depth, clinical attachment loss, and radiographic bone loss
  Interventions: Other: Collection of PICF samples
- Peri-implant Health: Peri-implant health is characterized by the absence of bleeding on probing, erythema, swelling, and suppuration in the peri-implant region
  Interventions: Other: Collection of PICF samples

INTERVENTIONS:
Other: Collection of PICF samples — TREM-1, MMP-8 and TIPM-1 levels reseach in PICF samples

SUMMARY:
The aim of this study was to evaluate the relationship between Triggering Receptor Expressed on Myeloid Cells-1 (TREM-1), Matrix Metalloproteinases-8 (MMP-8) and Tissue Inhibitors of Metalloproteinases-1 (TIMP-1) levels in peri-implant crevicular fluid (PICF) in peri-implantitis patients.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the relationship between TREM-1, MMP-8 and TIMP-1 levels in peri-implant crevicular fluid (PICF) in patients with peri-implantitis, and the correlation of these markers with clinical periodontal parameters.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy
* Pregnancy or lactation

Exclusion Criteria:

* osteoporosis
* rheumatoid arthritis
* autoimmune disease
* diabetes

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients had at least one implant, and this implant had been in place for at least one year since the implant-supported prosthesis was made.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2023-06-01 (Actual); Primary Completion 2023-12-15 (Actual); Study Completion 2024-05-20 (Actual)

PRIMARY OUTCOMES:
TREM-1, MMP-8 and TIMP-1 levels in PICF samples | 1 month
  TREM-1, MMP-8, and TIMP-1 levels in PICF samples were measured by ELISA method

CONTACTS AND LOCATIONS:
Locations (1):
- Aydın Adnan Menderes University, Aydin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided